CLINICAL TRIAL: NCT06488365
Title: In Vivo Liquid Biopsy for Early Detection of Metastatic Melanoma
Brief Title: In Vivo Liquid Biopsy of Melanoma (Cytophone)
Acronym: Cytophone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cytoastra (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00075507
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Melanoma; Circulating Tumor Cells; Metastatic Melanoma; Diagnosis
Keywords: melanoma; circulating tumor cells (CTCs); in vivo liquid biopsy; metastasis; diagnosis and prognosis
MeSH Terms: conditions — Melanoma; Neoplastic Cells, Circulating; Disease; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Healthy subjects and melanoma patients will be tested in this study. All subjects will receive the same Cytophone intervention (testing). Healthy subjects will receive one Cytophone test, and melanoma patients will receive four tests. There will be four cohorts to the study:
  Cohort 1: 30 healthy subjects to address the calibration purpose. Cohort 2: 50 stage 0-I melanoma patients to link the presence of CTCs in blood circulation or increase in CTC count with metastatic disease initiation.
  Cohort 3: 50 stage II melanoma patients to define the correlation between CTC count and metastatic disease initiation/progression and further recurrence.
  Cohort 4: 50 stage III-IV melanoma patients to link CTC counts, metastatic disease progression and therapy efficiency.
Masking Description: All study participants will be blinded from their results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cytophone application (Experimental): It is anticipated that Cytophone diagnostic procedure will start with 30-min preparation including ultrasound imaging of an examined vessel, photo of a skin area above the vessel and quick navigation of the PAFC probe on the vessel using near-infrared viewer. After completion, the Cytophone monitoring will be conducted for 30-60 min and will include noninvasive irradiation of the vessel by a laser beam(s) using a safe for human laser energy level.
  Interventions: Device: Cytophone

INTERVENTIONS:
Device: Cytophone — The Cytophone clinical prototype incorporates two pulse lasers, optical system for delivery of laser light to the skin, ultrasound transducer array and detection electronics for acquisition of acoustic waves from CTCs.
  Parameters of lasers:
  C-Wedge 1064 (Bright Solutions, Cura Carpignano (PV), Italy): Wavelength,1064 nm; pulse width, 0.6 ns; pulse rate: 1 kHz; pulse energy, 240 μJ.
  C-Wedge 18901 (Bright Solutions, Cura Carpignano (PV), Italy):
  Wavelength, 770 nm; pulse width 3 ns; pulse rate, 1 kHz; pulse energy, 240 μJ. Detection of acoustic waves from CTCs is performing by a focused ultrasound transducer array placed in an acoustic contact with the skin of the subject with ultrasound gel. The signals from the transducers are amplified with a 16 channel amplifier, then digitized by a 12-bit, 500 MSPS high speed board digitizer (ATS9350, AlazarTech, Canada). This information is then transferred to a data recording system using a secure computer.
  Other Names: Photoacoustiv flow cytometry (PAFC) in vivo

SUMMARY:
The Cytophone is a first in the world patented system to identify and count single circulating melanoma cells in blood circulation inside the human body. The Cytophone has a unique capability to find rare melanoma cells in the blood by an assessment of 100-500 times greater amounts of blood volume than routine blood tests. The important benefit of the Cytophone diagnosis is that the test does not require injection or any skin incision (i.e., non-invasiveness). The goal of this clinical trial is to demonstrate evidence of the capability of the Cytophone test to indicate a risk of metastasis and define CTC counts that correlate with melanoma recurrence, progression of metastatic disease, and therapy efficacy. The investigators believe that clinical trials will provide evidence that the Cytophone can diagnose risk of melanoma metastasis and recurrence earlier than existing methods.

DETAILED DESCRIPTION:
The majority of melanoma deaths are associated with metastasis that are formed by cancer cells shedding from the primary tumor that enter the circulation and spread to distant organs via blood circulation. These cells in blood are referred to as circulating tumor cells (CTCs). Growing evidence suggests that metastasis is an early event in melanoma patients, often occurring before metastases are clinically detectable. Therefore, detection of CTCs using liquid biopsy assays should be considered as an effective tool to diagnose early the risk of metastasis progression. Taking into account the link of CTCs with metastasis, CTCs have an advantage over many other biomarkers in identifying patients for early therapeutic intervention at a stage when the disease is still manageable and possibly curable. Overall, CTCs are in the blood circulation in early stage disease, yet they are typically detected in later stage disease. Currently, the main issue restricting the use of CTCs for early melanoma detection relates to the low sensitivity of existing assays due to assessment of limited blood volume (i.e., blood samples in vitro). To maximize the blood volume available for analysis, in vivo CTC enumeration without labelling in a large blood volume using the Cytophone device was developed by our team. The Cytophone represents a photoacoustic (PA) flow cytometry (PAFC) diagnostic platform. Our feasibility clinical study has demonstrated the detection of CTCs in 49 of 50 melanoma patients (sensitivity 98%) and in 0 of 18 in healthy subjects (control group). The investigators received clinical evidence of the Cytophone's capability to diagnose 0.001 CTCs/mL which is significantly higher than sensitivity of existing testing methodologies. This threshold of the sensitivity is 130-times better than the sensitivity of the in vitro CellSearch (Menarini) assay which is only assay approved by FDA for clinical testing of CTCs (1 CTC in 7.5 mL; 0.13 CTCs/mL).

The Goal of this clinical study is to determine whether the Cytophone can be used for in vivo detection and enumeration of circulating tumor cells (CTCs) in the melanoma patients at different disease stages with focus on early diagnosis, early assessment of disease recurrence and monitoring of therapy efficiency. It is expected that the detection limit of CTCs will be improved at least an order of magnitude compared to the detection limits of existing methods. The test results are intended to use in conjunction with other clinical diagnostic methods.

The investigators hypothesize that our CTC assay, in vivo, provides earlier, rapid and more accurate diagnosis and prognosis of metastasis progression in melanoma patients. To achieve our goal, the investigators will accomplish the following primary and secondary objectives:

The primary objectives:

1. Obtain evidence that a positive Cytophone CTC test indicates a risk of metastasis development.
2. Define thresholds of CTC counts that correlate with melanoma recurrence and progression of metastatic disease.

The secondary objective:

1. Determine if the Cytophone diagnoses the risk of melanoma metastasis progression and recurrence earlier than existing methods.

ELIGIBILITY:
Inclusion Criteria:

* Histological documented diagnosis of melanoma;
* Participants having provided informed consent with signature on informed consent form: the informed consent process should be complete with full discussion of all requirements and possible risks;
* Must be able to sit for up to 60 minutes.

Exclusion Criteria:

* Unable to provide informed consent to participate in the study, such as a mental condition rendering the participant unable to understand the nature, scope, and possible consequences of the study;
* Clinically relevant cardiovascular, hepatic, neurological (e.g., evidence of organic brain syndrome), endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the participant at risk by participating in the study;
* Persistent significant or severe infection, either acute or chronic;
* Pregnant or breast-feeding women or those who plan to become pregnant during the study;
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy;
* Any known history of severe preexisting constipation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Identify and count CTCs in blood in vivo | nine months
  Link CTC counts with early melanoma progression and recurrence efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Galanzha, PhD, Study Director — Cytoastra
Locations (1):
- SSM Health Dean Medical Group Specialty Services, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galanzha EI, Shashkov EV, Spring PM, Suen JY, Zharov VP. In vivo, noninvasive, label-free detection and eradication of circulating metastatic melanoma cells using two-color photoacoustic flow cytometry with a diode laser. Cancer Res. 2009 Oct 15;69(20):7926-34. doi: 10.1158/0008-5472.CAN-08-4900. Epub 2009 Oct 13. PMID 19826056
- [Background] Galanzha EI, Zharov VP. Circulating Tumor Cell Detection and Capture by Photoacoustic Flow Cytometry in Vivo and ex Vivo. Cancers (Basel). 2013 Dec 10;5(4):1691-738. doi: 10.3390/cancers5041691. PMID 24335964
- [Result] Galanzha EI, Menyaev YA, Yadem AC, Sarimollaoglu M, Juratli MA, Nedosekin DA, Foster SR, Jamshidi-Parsian A, Siegel ER, Makhoul I, Hutchins LF, Suen JY, Zharov VP. In vivo liquid biopsy using Cytophone platform for photoacoustic detection of circulating tumor cells in patients with melanoma. Sci Transl Med. 2019 Jun 12;11(496):eaat5857. doi: 10.1126/scitranslmed.aat5857. PMID 31189720

DOCUMENTS (2):
  • Study Protocol (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT06488365/Prot_000.pdf
  • Informed Consent Form (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT06488365/ICF_001.pdf